CLINICAL TRIAL: NCT01242488
Title: Randomized, Double-blind, Placebo-controlled, Dose Ranging Study With an Active Comparator to Evaluate the Efficacy and Safety of CDP6038 Administered Subcutaneously for 12 Weeks to Subjects With Rheumatoid Arthritis Having Previously Failed TNF-blocker Therapy
Brief Title: Efficacy and Safety of CDP6038 in Patients With Rheumatoid Arthritis With an Unsuccessful Response to Anti-Tumor Necrosis Factor (Anti-TNF) Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UCB Pharma (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: RA0056; 2010-020839-39 (EudraCT Number)
Record Dates: First submitted 2010-11-15; First posted 2010-11-17 (Estimated); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid Arthritis; CDP6038; Interleukin-6; Tocilizumab
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — olokizumab; tocilizumab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (9):
- CDP6038 60 mg sc every 2 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo iv
- CDP6038 60 mg sc every 4 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo sc; Other: Placebo iv
- CDP6038 120 mg sc every 2 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo iv
- CDP6038 120 mg sc every 4 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo sc; Other: Placebo iv
- CDP6038 240 mg sc every 2 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo iv
- CDP6038 240 mg sc every 4 weeks plus methotrexate (Experimental)
  Interventions: Biological: CDP6038; Other: Placebo sc; Other: Placebo iv
- Tocilizumab 8 mg/kg iv every 4 weeks plus methotrexate (Active Comparator)
  Interventions: Biological: Tocilizumab (Actemra or RoActemra); Other: Placebo sc
- Placebo sc every 2 weeks plus methotrexate (Placebo Comparator)
  Interventions: Other: Placebo sc; Other: Placebo iv
- Placebo sc every 4 weeks plus methotrexate (Placebo Comparator)
  Interventions: Other: Placebo sc; Other: Placebo iv

INTERVENTIONS:
Biological: CDP6038 — 60 mg subcutaneously (sc) at Weeks 0, 2, 4 6, 8, and 10
  Arms: CDP6038 60 mg sc every 2 weeks plus methotrexate
Biological: CDP6038 — 120 mg sc at Weeks 0, 2, 4 6, 8, and 10
  Arms: CDP6038 120 mg sc every 2 weeks plus methotrexate
Biological: CDP6038 — 240 mg sc at Weeks 0, 2, 4 6, 8, and 10
  Arms: CDP6038 240 mg sc every 2 weeks plus methotrexate
Biological: Tocilizumab (Actemra or RoActemra) — 8 mg/kg intravenously (iv) at Weeks 0, 4 and 8
  Arms: Tocilizumab 8 mg/kg iv every 4 weeks plus methotrexate
Biological: CDP6038 — 60 mg sc at Weeks 0, 4 and 8
  Arms: CDP6038 60 mg sc every 4 weeks plus methotrexate
Biological: CDP6038 — 240 mg sc at Weeks 0, 4 and 8
  Arms: CDP6038 240 mg sc every 4 weeks plus methotrexate
Biological: CDP6038 — 120 mg sc at Weeks 0, 4 and 8
  Arms: CDP6038 120 mg sc every 4 weeks plus methotrexate
Other: Placebo sc — 0.9% Sodium chloride for injection at Weeks 0, 2, 4 6, 8, and 10
  Arms: Placebo sc every 2 weeks plus methotrexate; Placebo sc every 4 weeks plus methotrexate; Tocilizumab 8 mg/kg iv every 4 weeks plus methotrexate
Other: Placebo sc — 0.9% Sodium chloride for injection at Weeks 2, 6 and 10
  Arms: CDP6038 120 mg sc every 4 weeks plus methotrexate; CDP6038 240 mg sc every 4 weeks plus methotrexate; CDP6038 60 mg sc every 4 weeks plus methotrexate
Other: Placebo iv — 0.9% Sodium chloride for injection at Weeks 0, 4 and 8
  Arms: CDP6038 120 mg sc every 2 weeks plus methotrexate; CDP6038 120 mg sc every 4 weeks plus methotrexate; CDP6038 240 mg sc every 2 weeks plus methotrexate; CDP6038 240 mg sc every 4 weeks plus methotrexate; CDP6038 60 mg sc every 2 weeks plus methotrexate; CDP6038 60 mg sc every 4 weeks plus methotrexate; Placebo sc every 2 weeks plus methotrexate; Placebo sc every 4 weeks plus methotrexate

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, pharmacokinetics, and immunogenicity of CDP6038 treatment in adult subjects with active rheumatoid arthritis who have had an inadequate response to anti-tumor necrosis factor (anti-TNF) therapy.

DETAILED DESCRIPTION:
CDP6038 is a protein (antibody) that blocks interleukin-6 (IL-6), a substance involved in the inflammation associated with rheumatoid arthritis. This is a multicenter, 12-week, randomized, double-blind, placebo- and active- controlled study comparing several doses and dosage regimens (every 2 weeks and every 4 weeks) of CDP6038 to placebo and tocilizumab in patients with active rheumatoid arthritis who have had an unsuccessful response to methotrexate and previous anti-TNF therapy. The study will test if CDP6038 is more efficacious than placebo in reducing the signs and symptoms of rheumatoid arthritis at 12 weeks while maintaining an adequate safety profile. In order to maintain the study blinding all subjects will be given a subcutaneous (sc) injection (under the skin) every 2 weeks, as well as an intravenous (iv) infusion every 4 weeks. In addition subjects must remain on stable weekly doses of methotrexate. Assessments during the study include evaluations of joint pain and swelling, laboratory blood and urine tests, physical examinations, vital signs, electrocardiograms, and questionnaires. Subjects who complete the 12-week study will be eligible to enroll in a long-term extension study receiving CDP6038.

ELIGIBILITY:
Inclusion Criteria:

* Have a diagnosis of rheumatoid arthritis (according to the 1987 ACR classification criteria OR a score of ≥6 as defined by the ACR/European League Against Rheumatism Classification and Diagnostic Criteria for rheumatoid arthritis ) for at least 6 months prior to screening
* Must have been treated with MTX 12.5-25 mg/week, for at least 6 weeks prior to screening. Doses of 10 to < 12.5mg/week are allowed if there is documented intolerance
* Have moderately to severely active rheumatoid arthritis disease with at least 6 tender and 6 swollen joints
* CRP ≥1.2 times the upper limit of normal (central laboratory) or erythrocyte sedimentation rate of more than 28mm/hour
* Intolerant or inadequate response to treatment (ie, TNF blocker failure)≥1 licensed TNF-blocker therapies within 2 years of screening

Exclusion Criteria:

* Have a diagnosis of any other inflammatory arthritis or secondary, noninflammatory type of arthritis, such as psoriatic arthritis, lupus, gout, or ankylosing spondylitis
* Wheelchair bound or bedridden.
* Disease modifying antirheumatic drugs (DMARDs) other than MTX.
* Treatment with tocilizumab or any other anti-IL-6 investigational therapies at any time.
* Treatment with other biologics within 4-24 weeks (depending on the biologic)
* History of ongoing, chronic or recurrent infections or recent serious or life-threatening infection
* Known concurrent acute or chronic viral hepatitis B or C infection or human immunodeficiency virus (HIV) infection.
* Vaccinations (other than injectable influenza or pneumococcal) within 8 weeks prior to screening or plan to receive vaccines during the study
* Concurrent or history of malignancy with the exception of nonmelanoma skin cancer successfully treated more than 2 years prior to screening or cervical cancer successfully treated more than 5 years prior to screening.
* History of chronic alcohol abuse or drug addiction within the last 1 year or current drug addiction or use of illicit drugs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 221 (Actual)
Dates: Start 2010-11; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in the Disease Activity Score (C-reactive protein) [DAS28(CRP)] for CDP6038 and placebo | Baseline, Week 12

SECONDARY OUTCOMES:
American College of Rheumatology 20% response (ACR20) rates for the CDP6038 and placebo arms. | From Baseline to Week 12
American College of Rheumatology 50% response (ACR50) rates for the CDP6038 and placebo arms. | From Baseline to Week 12
American College of Rheumatology 70% response (ACR70) rates for the CDP6038 and placebo arms. | From Baseline to Week 12

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call Center, Study Director — +1 877 822 9493 (UCB)
Locations (82):
- United States (74):
  - 166, Mesa, Arizona
  - 154, Paradise Valley, Arizona
  - 118, Scottsdale, Arizona
  - 103, Hot Springs, Arkansas
  - 125, Jonesboro, Arkansas
  - 127, Covina, California
  - 148, La Jolla, California
  - 184, Long Beach, California
  - 177, Los Angeles, California
  - 104, Palo Alto, California
  - 149, Sacramento, California
  - 158, San Diego, California
  - 129, Santa Maria, California
  - 164, Upland, California
  - 107, Wildomar, California
  - 141, Hamden, Connecticut
  - 137, Norwalk, Connecticut
  - 101, Trumbull, Connecticut
  - 111, Lewes, Delaware
  - 176, Aventura, Florida
  - 186, Daytona Beach, Florida
  - 151, DeBary, Florida
  - 114, Jupiter, Florida
  - 183, Pinellas Park, Florida
  - 178, Sarasota, Florida
  - 140, South Miami, Florida
  - 157, Tampa, Florida
  - 130, Gainesville, Georgia
  - 162, Newnan, Georgia
  - 153, Savannah, Georgia
  - 113, Stockbridge, Georgia
  - 116, Idaho Falls, Idaho
  - 160, Moline, Illinois
  - 156, Rock Island, Illinois
  - 168, Springfield, Illinois
  - 133, Cedar Rapids, Iowa
  - 172, Kansas City, Kansas
  - 185, Saint Clair Shores, Michigan
  - 112, St Louis, Missouri
  - 134, St Louis, Missouri
  - 102, Lincoln, Nebraska
  - 171, Freehold, New Jersey
  - 163, New Brunswick, New Jersey
  - 152, Toms River, New Jersey
  - 174, Brooklyn, New York
  - 115, Rochester, New York
  - 109, Belmont, North Carolina
  - 170, Charlotte, North Carolina
  - 150, Cincinnati, Ohio
  - 108, Columbus, Ohio
  - 100, Dayton, Ohio
  - 110, Oklahoma City, Oklahoma
  - 165, Duncansville, Pennsylvania
  - 117, Wexford, Pennsylvania
  - 105, Nashville, Tennessee
  - 106, Nashville, Tennessee
  - 120, Amarillo, Texas
  - 135, Austin, Texas
  - 128, Dallas, Texas
  - 126, Houston, Texas
  - 132, Houston, Texas
  - 138, Houston, Texas
  - 181, Houston, Texas
  - 145, Mesquite, Texas
  - 143, Nassau Bay, Texas
  - 122, San Antonio, Texas
  - 144, Tomball, Texas
  - 142, Victoria, Texas
  - 121, Salt Lake City, Utah
  - 139, Chesapeake, Virginia
  - 119, Seattle, Washington
  - 175, Tacoma, Washington
  - 136, Beckley, West Virginia
  - 167, Clarksburg, West Virginia
- Belgium (2):
  - 401, Brussels
  - 400, Liège
- United Kingdom (6):
  - 209, Torquay, Devon
  - 201, Wigan, Lancashire
  - 206, Essex
  - 205, London
  - 204, Newcastle upon Tyne
  - 208, Southampton

REFERENCES:
- [Derived] Genovese MC, Fleischmann R, Furst D, Janssen N, Carter J, Dasgupta B, Bryson J, Duncan B, Zhu W, Pitzalis C, Durez P, Kretsos K. Efficacy and safety of olokizumab in patients with rheumatoid arthritis with an inadequate response to TNF inhibitor therapy: outcomes of a randomised Phase IIb study. Ann Rheum Dis. 2014 Sep;73(9):1607-15. doi: 10.1136/annrheumdis-2013-204760. Epub 2014 Mar 18. PMID 24641941